CLINICAL TRIAL: NCT06642025
Title: An Open-label, Single-arm Clinical Study of EX02 CAR-T Therapy for Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: EX02 CAR-T Cells for Relapsed and Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhimin Zhai (Other)
Collaborators: Zeno Therapeutics Pte. Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Zhimin Zhai, Chief of Hematology Department, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024-001(F1)
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia (AML); CAR-T
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Cell Injection (Experimental)
  Interventions: Biological: CAR-T Cell Injection

INTERVENTIONS:
Biological: CAR-T Cell Injection — Conditioning chemotherapy: Lymphodepletion regimen consisting of fludarabine 25 mg/m2/day and cyclophosphamide 250 mg/m2/day for 3 consecutive days, administered 48 hours before intraperitoneal infusion.
  On the day of administration, premedication with 500mg of acetaminophen orally and 20mg of promethazine intramuscularly or intravenously (or other non-steroidal anti-inflammatory drugs and antihistamines) should be given 30 minutes before intraperitoneal infusion.
  The therapeutic dose of CAR-T cells is defined as intravenous injection of 1.0E6 CAR-T cells/kg as the initial standard dosage.

SUMMARY:
This is a early Phase 1 open-label, single-arm clinical study of EX02 CAR-T therapy for relapsed and refractory acute myeloid leukemia.

Each participant will undergo leukapheresis after enrolment, receive treatment of the conditioning chemotherapy of cyclophosphamide and fludarabine, and an an intravenous infusion of CAR-T cells.

Each participant will proceed through the following study procedures:

* Screening
* Enrollment/Leukapheresis
* Conditioning chemotherapy
* CAR T treatment
* Post-treatment assessment
* Long-term follow-up

ELIGIBILITY:
Inclusion Criteria:

1. According to the Chinese Adult Acute Myeloid Leukemia (AML) Diagnosis and Treatment Guidelines (2023 edition/previous edition), patients diagnosed with acute myeloid leukemia (AML) and meeting the diagnostic criteria for refractory AML are eligible, including: initial treatment cases with no response after two courses of standard therapy; relapse within 12 months after achieving complete remission (CR) and failure of consolidation therapy; relapse after 12 months with no response to conventional chemotherapy; two or more relapses; and presence of extramedullary leukemia.
2. Peripheral blood, bone marrow, or extramedullary lesion specimens showing leukemia cells with positive surface expression of EX02;
3. ECOG performance status score of 0-2;
4. Age ≥18 and ≤70 years, any gender;
5. Blood cell examination meeting the following conditions: hemoglobin > 60g/L, normal T lymphocyte count (CD3+) > 0.5×10^9/L, platelet count > 30×10^9/L;
6. Negative pregnancy test for women of childbearing potential before the start of the trial, and agreement to use effective contraception measures during the trial until the final follow-up; male participants of reproductive potential agreeing to use effective contraception measures during the trial until the final follow-up;
7. Voluntary participation in this clinical study: after fully understanding the study content, voluntary signing of the informed consent form, and commitment to complete all trial procedures and activities.

Exclusion Criteria:

1. Active hepatitis A, B, C, HIV infection, or other severe active infections that are not yet controlled;
2. History of acquired immune deficiency syndrome (AIDS) or long-term use of immunosuppressants due to other diseases (including steroids, equivalent to prednisone >15mg/day);
3. Conditions of the heart function: a. New York Heart Association (NYHA) class III or IV heart failure; b. Myocardial infarction or coronary artery bypass surgery within the six months prior to enrollment; c. Clinically significant ventricular arrhythmia or unexplained syncope; d. History of severe non-ischemic cardiomyopathy; e. History of cardiac dysfunction (left ventricular ejection fraction <45%) within 8 weeks before enrollment;
4. Pregnant or lactating women; participants (both male and female) unwilling to use contraception;
5. Severe liver or kidney dysfunction: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels exceeding 3 times the upper limit of normal, bilirubin exceeding 3 times the upper limit of normal; serum creatinine ≥ 178 μmol/L (decompensated phase);
6. History of severe allergic reactions to any drugs planned for use in this study;
7. Recipients of hematopoietic stem cell transplantation must have discontinued immunosuppressants for at least 6 weeks before enrollment and have no signs of graft-versus-host disease;
8. Other conditions deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAE) | From the infusion (Day 0) to 3 months
  TEAE is defined as any adverse event that occurs within 90 days after the first injection of EX02 CAR-T, or that existed before treatment and worsened after treatment. All adverse events are graded according to CTCAE v4.0, classified, and then the incidence rate is calculated. In addition, according to the definition of this study, the occurrence of CAR-T cell therapy-specific CRS and ICANS, as well as their grading, management, and prognosis are evaluated, and the incidence rates are calculated separately, with specific patient details recorded.
Overall Response Rate (ORR) | From the infusion (Day 0) to Day 60
  Overall response rate=number of complete remission(CR) (including incomplete hematologic recovery (CRi)) + number of partial remission (PR) / total number of treated cases, determined by the investigator according to the 2023 Chinese Diagnosis and Treatment Guidelines for Adult Acute Myeloid Leukemia (non-acute promyelocytic leukemia).

SECONDARY OUTCOMES:
PFS | 12 months
  The time from the onset of leukocyte apheresis to the appearance of tumor progression or death
OS | 12 months
  OS, The time between leukocyte apheresis and death from any cause
ECOG scoring | 2 months
  Zubrod-ECOG-WHO method for assessing and comparing the physical status of patients before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No